CLINICAL TRIAL: NCT03207932
Title: Ultrasound Guidance Versus Anatomical Landmarks for Succlavic and Femoral Vein Catheterisation: an Observational Prospective Study
Brief Title: Ultrasound Guidance Versus Anatomical Landmarks for CVC Catheterisation:
Status: Completed | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Francesco Forfori, Professor, University of Pisa
Other Study IDs: UPisa - subclavian/femoral
Record Dates: First submitted 2017-07-02; First posted 2017-07-05 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Success Rate for Subclavian or Femoral Vein Catetherisation
MeSH Terms: interventions — Catheterization, Central Venous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ultrasound: CVC insertion using ultrasound
  Interventions: Procedure: Central vein catheterisation
- landmark technique: CVC insertion using landmark technique
  Interventions: Procedure: Central vein catheterisation

INTERVENTIONS:
Procedure: Central vein catheterisation — ultrasound guided versus landmark central vein catheterisation

SUMMARY:
anatomical landmarks on the body surface were used to insert central vein catheter. However, ultrasound technique is emerging as a new technique for vein catheterisation. For subclavian and femoral vein catheterisation, up to now, there is a lack of evidence of the superiority of one technique over the other.

ELIGIBILITY:
Inclusion Criteria:

* patients needing CVC

Exclusion Criteria:

* refusal of consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: intensive care patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
The success rate for succlavic or femoral vein catetherisation using ultrasound versus landmark technique at the first attempt | during catheterization procedure
  success rate

CONTACTS AND LOCATIONS:
Locations (1):
- Francesco Forfori, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No